CLINICAL TRIAL: NCT00039000
Title: A Phase III Study of Heat Shock Protein-Peptide Complex (HSPPC-96) Versus Physician's Choice Including Interleukin-2 and/or Dacarbazine/Temozolomide-based Therapy and/or Complete Tumor Resection in Stage IV Melanoma
Brief Title: Study of Heat Shock Protein-Peptide Complex (HSPPC-96) Versus IL-2/DTIC for Stage IV Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-100-21; NCT00047359 (obsolete NCT alias)
Record Dates: First submitted 2002-06-06; First posted 2002-06-10 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Malignant Melanoma
Keywords: Immunotherapy, Cancer, Melanoma, Skin Cancer, tumor
MeSH Terms: conditions — Melanoma; Neoplasms; Skin Neoplasms | interventions — vitespin

INTERVENTIONS:
Drug: HSPPC-96 or Oncophage

SUMMARY:
The primary goal of this study is to determine if people with metastatic melanoma who receive Heat Shock Protein-Peptide Complex - 96 (HSPPC-96 or Oncophage) after surgery live longer than people who may or may not have surgery but who receive conventional chemotherapy including IL-2/DTIC. A second goal is to determine the safety and frequency of side effects in subjects who receive therapy with HSPPC-96.

DETAILED DESCRIPTION:
Primary Objective:

* To determine whether subjects with stage IV melanoma randomized to HSPPC-96 have longer survival than subjects randomized to physician's choice including interleukin-2 and/or dacarbazine/temozolomide and/or complete tumor resection.

Secondary Objective:

* To determine frequency of adverse events in subjects randomized to HSPPC-96.

ELIGIBILITY:
Eligibility Assessment:

(The following assessments must be obtained within three weeks prior to randomization into the study)

* Medical history and physical examination (including EGOG score, evidence of immunosuppression);
* CT/MRI of the chest, abdomen and pelvis;
* Clinical examination;
* CT/MRI of the brain;
* Complete Blood Count with differential including platelets;
* Electrolytes (Na, Cl, K, HCO3, Ca, Mg, PO4);
* Renal function tests (BUN and creatinine);
* Liver function tests (bilirubin, AST, ALT);
* Serum pregnancy test for all women of childbearing potential.

Inclusion Criteria:

* Stage IV Melanoma (AJCC);
* No prior therapy for stage IV melanoma;
* No prior therapy with interleukin-2 and/or dacarbazine/temozolomide within the past 12 months prior to study entry;
* Candidate for surgical resection of some/all sites of melanoma and expected to obtain greater tan or equal to 7 grams of viable cancer tissue (in aggregate), which is equivalent to a greater than or equal to 2 cm lesion on CT/MRI or clinical examination;
* No brain metastases;
* ECOG score 0 or 1;
* Adequate cardiac function;
* Adequate hematopoietic, liver and renal function;
* Female subjects of child-bearing potential must agree to use contraception during the study
* Signed written informed consent.

Exclusion Criteria:

* Mucosal or ocular melanomas;
* Other malignancies treated within the last five years, except in situ cervix carcinoma or non-melanoma skin cancer;
* Primary or secondary immunodeficiency, in the opinion of the investigator (including immunosuppressive disease, or use of systemic corticosteroids or other immunosuppressive medications);
* Prior splenectomy;
* Uncontrolled infection or other serious medical illnesses;
* Women who are pregnant or breast-feeding;
* Subjects participating in any other studies requiring administration of an investigational drug/biologic agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2002-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (77):
- United States (35):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Berkeley, California
  - Los Angeles, California
  - Stanford, California
  - Vista, California
  - Denver, Colorado
  - Farmington, Connecticut
  - Jacksonville, Florida
  - Lakeland, Florida
  - Miami Beach, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Columbia, Missouri
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - New Brunswick, New Jersey
  - New York, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Knoxville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Madison, Wisconsin
- Australia (5):
  - Adelaide
  - Camperdown
  - Melbourne
  - Newcastle
  - Wentworthville
- Hungary (4):
  - Budapest
  - Debrecen
  - Pécs
  - Szeged
- Italy (4):
  - Aviano
  - Genova
  - Milan
  - Rimini
- Poland (3):
  - Bialystock
  - Bydgoszcz
  - Krakow
- Russia (11):
  - Arkhangelsk
  - Chelyabinsk
  - Kazan'
  - Krasnodar
  - Moscow
  - Novosibirsk
  - Ryazan
  - Saint Petersburg
  - Samara
  - Stavropol
  - Voronezh
- Sweden (3):
  - Gothenburg
  - Lund
  - Vaxjo
- Ukraine (9):
  - Dnipro
  - Donetsk
  - Ivano-Frankivsk
  - Kiev
  - Kryvyi Rih
  - Lviv
  - Odesa
  - Uzhhorod
  - Vinnitsa
- United Kingdom (3):
  - Leeds
  - London
  - Manchester